CLINICAL TRIAL: NCT00542958
Title: A Phase I Dose-escalation Study of NK012 Administered Intravenously as a Single Dose Every Three Weeks in Patients With Refractory Solid Tumors
Brief Title: Study of NK012 in Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: N06-10089
Record Dates: First submitted 2007-10-11; First posted 2007-10-12 (Estimated); Last update posted 2019-10-28 (Actual); Status verified 2013-03

CONDITIONS: Cancer
Keywords: Cancer; Refractory solid tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NK012 (Experimental): This is a Phase I dose-escalation study of the intravenous administration of NK012 in patients with refractory solid tumors. Patients will receive NK012 as an intravenous infusion over 30 minutes on Day 1 followed by a 20-day observation period for a total of 21 days (3 weeks) per cycle. Two patient populations will be evaluated separately: patients with UGT1A1*28 genotype homozygous wild type (wt/wt) and heterozygous (wt/*28) variants as one group, and patients with UGT1A1*28 homozygous variant (*28/*28) as another group. Dose-escalation in each patient population will proceed according to the predefined dose level.
  For UGT1A1*28 (wt/wt and wt/*28) patients, at least 3 evaluable patients will be treated at each dose level.
  UGT1A1 homozygous (*28/*28) patients will be treated at 50% of the current dose level.
  Patients will receive up to 6 cycles of NK012, unless they experience unacceptable toxicity or disease progression, requiring withdrawal from the study.
  Interventions: Drug: NK012

INTERVENTIONS:
Drug: NK012 — 9.0, 12.0, 16.0, 21.0, 28.0 mg/m^2, and to be determined. Intravenous infusion

SUMMARY:
The purpose of this study is to determine whether NK012 is safe and effective in the treatment of refractory solid tumors

DETAILED DESCRIPTION:
This is a Phase I dose-escalation study of the intravenous administration of NK012 in patients with refractory solid tumors. Patients will receive NK012 as an intravenous infusion over 30 minutes on Day 1 followed by a 20-day observation period for a total of 21 days (3 weeks) per cycle. Two patient populations will be evaluated separately: patients with UGT1A1*28 genotype homozygous wild type (wt/wt) and heterozygous (wt/*28) variants as one group, and patients with UGT1A1*28 homozygous variant (*28/*28) as another group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant solid tumor for which there are no known regimens or protocol treatments of higher efficacy or priority
* Failed conventional therapy for the cancer or have a malignancy for which a conventional therapy does not exist
* Recovered from all acute adverse effects of prior therapies, excluding alopecia (hair loss)
* Life expectancy of at least 12 weeks and an EOCG performance status of 0 or 1
* 18 years of age or older
* Adequate kidney, liver, and bone marrow function
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or have not recovered from adverse effects due to agents administered more than 4 weeks earlier
* Receiving any other investigational agent
* History of brain metastases or spinal cord compression, unless irradiated a minimum of 4 weeks before study entry and stable without requirement for corticosteroids for > 1 week
* History of allergic reactions attributed to compounds of similar chemical composition to NK012
* Concurrent serious infections (i.e., requiring an intravenous antibiotic)
* Pregnant women or women of childbearing potential who are not using methods to avoid pregnancy; a negative pregnancy test (urine or serum) must be documented at baseline and before every NK012 administration for women of childbearing potential; no breast-feeding while on study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris or psychiatric illness/social situations that would limit compliance with study requirements
* Significant cardiac disease
* History of serious ventricular arrhythmia
* Positive for anti-HbsAg, anti-HCV, anti-HIV, or anti-syphilis antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-03; Primary Completion 2008-04 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity of NK012 in patients with UGT1A1*28 (wt/wt and wt/*28) genotype | At the end of Cycle 1 (each cycle is 21 days)
Maximum tolerated dose of NK012 in patients with UGT1A1*28 (wt/wt and wt/*28) genotype | At the end of Cycle 1 (each cycle is 21 days)
Recommended phase II dose of NK012 in patients with UGT1A1*28 (wt/wt and wt/*28) genotype | At the end of Cycle 1 (each cycle is 28 days)
  After MTD was determined, the administration schedule was changed to every 28 days per cycle, considering patient safety.

SECONDARY OUTCOMES:
Toxicity profile of NK012 in all patients | Through study completion (6 cycles of study drug administration period and 30 days of follow-up period), an average of 5 months for 21-day cycle or 6 months for 28-days cycle.
Antitumor activity of NK012 according to RECIST criteria in all patients | Through study completion (6 cycles of study drug administration period and 30 days of follow-up period), an average of 5 months for 21-day cycle or 6 months for 28-days cycle.
  Overall response will be evaluated every 2 cycles
Pharmacokinetic parameter: Maximum concentration (Cmax) | Sampling during Cycle 1 (first 3 weeks) and up to Day 3 of Cycle 2, if applicable, total 24 days for 21-days cycle or 31 days for 28-day cycle.
Pharmacokinetic parameter: Time to reach the maximum concentration (Tmax) | Sampling during Cycle 1 (first 3 weeks) and up to Day 3 of Cycle 2, if applicable, total 24 days for 21-days cycle or 31 days for 28-day cycle.
Pharmacokinetic parameter: Terminal-phase half life (T1/2z) | Sampling during Cycle 1 (first 3 weeks) and up to Day 3 of Cycle 2, if applicable, total 24 days for 21-days cycle or 31 days for 28-day cycle.
Pharmacokinetic parameter: Area under the concentration-time curve for time zero to infinity (AUCinf) | Sampling during Cycle 1 (first 3 weeks) and up to Day 3 of Cycle 2, if applicable, total 24 days for 21-days cycle or 31 days for 28-day cycle.
Pharmacokinetic parameter: Total body clearance (CLtot) | Sampling during Cycle 1 (first 3 weeks) and up to Day 3 of Cycle 2, if applicable, total 24 days for 21-days cycle or 31 days for 28-day cycle.
Pharmacokinetic parameter: Volume of distribution at steady-state (Vss) | Sampling during Cycle 1 (first 3 weeks) and up to Day 3 of Cycle 2, if applicable, total 24 days for 21-days cycle or 31 days for 28-day cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, III, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Sarah Cannon Research Institute, Nashville, Tennessee, United States